CLINICAL TRIAL: NCT04679428
Title: Immunological Characteristics of COVID-19 Patients and Determination of Neutralizing Antibodies Against SARS-CoV-2 Virus
Brief Title: Immunological Characteristics of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Collaborators: National Institute of Chemistry, Slovenia (Unknown)
Responsible Party: Principal Investigator, Peter Korošec, Assoc Prof Peter Korošec, BSc (Biol), PhD, The University Clinic of Pulmonary and Allergic Diseases Golnik
Other Study IDs: Golnik_Covid-19
Record Dates: First submitted 2020-12-21; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Covid-19; SARS-CoV-2; immunology; TBNK Cells; neutralizing antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will look at the immunological characteristics of COVID-19 patients and determine neutralizing antibodies against SARS-CoV-2 virus.

DETAILED DESCRIPTION:
The immunogram (quantitative TBNK immunophenotipisation) will be performed by flow cytometry, the antibody response will be determined by IVD ELISa.

Clinical biochemical and immunochemical (ECLIA) tests (including IL-6) will be performed on Cobas analyzers. Hemogram with differential blood picture will be performed with a hematology analyzer Sysmex XN 3100, examination of blood smears with CellaVision system or. microscope. Coagulation tests will be performed on BCS XP analyzers.

An in-house system for the analysis of SARS-CoV-2 virus fusion inhibitors on human cells will be used to detect the ability of antibodies from patients' serum to neutralize the virus and thus potential protection against re-infection. The system is quantitative, meaning that the titer of such antibodies could be determined, and thus the potential level of protection would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Provide written consent before being included in the essay.

Positive cases of COVID-19 (based on polymerase chain reaction or positive antigen test for SARS-CoV-2).

Exclusion Criteria:

Patients who are unable to give consent or who are unable to follow up will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients recruited at University Clinic of Pulmonary and Allergic Diseases Golnik.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-05-07 (Estimated); Study Completion 2023-05-07 (Estimated)

PRIMARY OUTCOMES:
Immunological changes during and after COVID-19 infection | July 2022
  Correlation between TBNK dynamic and increase of neutralising antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Peter Korošec, PhD, Principal Investigator — Head of the Laboratory for Clinical Immunology and Molecular Genetics
Locations (1):
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Slovenia